CLINICAL TRIAL: NCT01440153
Title: Influence of an Additional Intervention Targeting Physical Fitness, Endurance and Motor Control, on Physical Condition and Musculoskeletal Injuries in Contemporary Dancers
Brief Title: Additional Exercise Program in Professional Dancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College of Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UZA-DRCT-2011
Record Dates: First submitted 2011-08-23; First posted 2011-09-26 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Musculoskeletal Diseases
Keywords: Dance; Injury; Physical condition; Exercise
MeSH Terms: conditions — Musculoskeletal Diseases; Wounds and Injuries; Motor Activity | interventions — Functional Laterality; Educational Status; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Intervention (Experimental)
  Interventions: Other: Exercise Intervention
- passive intervention (Active Comparator)
  Interventions: Other: Passive Intervention

INTERVENTIONS:
Other: Exercise Intervention — Participants from group A receive an active program aiming at improving their cardiovascular endurance, muscular strength and motor control. The level for cardiovascular training is based on the results of the maximal exercise test performed during baseline assessment. The level of training is determined at a level of 70% of the predicted maximal heart rate and was increased every 6 weeks with 5%, ending at 85%. Heart rate will be monitored during the training.
  Other Names: Fitness; Motor control; Physical condition
  Arms: Active Intervention
Other: Passive Intervention — Participants from group B will receive an alternative program, in which all active parts are replaced by passive interventions. Several education sessions will be given regarding different topics, such as stress management, nutrition, injuries, etc. In addition, also practical sessions well be held to practice massage, passive stretching, taping.
  Other Names: stress management; education; taping; massage
  Arms: passive intervention

SUMMARY:
Professional dancing requires an almost perfect control of technical skills, combined with a good physical condition. To meet the demands of choreography, dancers need an adequate aerobic endurance capacity, muscular strength as well as flexibility and motor control (Twitchett et al. 2009; Roussel et al. 2009). One could compare these requirements to those of an athlete. In contrasts to athletes, only few attention has been given to the prevention of injuries in dancers. Professional dancers are at high risk to develop musculoskeletal injuries, especially, soft tissue and overuse injuries to lower extremities and spine(Hincapié et al, 2008). Several potential risk factors for injury have been suggested, such as a reduced level of aerobic fitness, lack of muscular strength, hypermobility of the joints and altered motor control of the lumbopelvic region but no conclusive evidence exists for any of these items separately.

Applying sports science principles to dance training may improve the performances of the dancers (Twitchett et al. 2009). Dancers demonstrate low aerobic fitness and muscle strength, in contrast to the high demands. Aerobic endurance of dancers is for example comparable to healthy adults with a sedentary life style.

Fitness programs, additional to regular dance classes, have only recently been considered (Twitchett et al. 2009). The advantages of additional training in athletes is beyond questioning. Nevertheless, this concept is relatively new for dancers. On the one hand, professional dancers do not consider themselves as a sportsmen but as artists (Wyon et al, 2007). On the other hand, choreographers and dancers fear the negative influence of training on body aesthetics.

Additional fitness training could improve physical fitness & motor control and may help with stress coping during public performances. Therefore, the purpose of this randomized controlled trial is to examine whether an additional intervention to regular dance lessons influences the physical condition and musculoskeletal injury rate in professional dancers.

DETAILED DESCRIPTION:
Prior to participation, all subjects receive verbal and written information addressing the nature of the study. First dancers are asked to fill in a self-established medical questionnaire, the Short Form 36 questionnaire (SF-36), the Dance Functional Outcome Scale (DFOS), the Baecke questionnaire, the Pain Catastrophizing Scale (PCS) and the Tampa Scale for Kinesiofobia (TSK). After a baseline assessment, consisting of an evaluation of the physical condition (maximal exercise test, evaluation of the respiratory capacity & evaluation of explosive muscle strength using a field test), a motor control evaluation of the lumbo-pelvic region and evaluation of anthropometric measurements, the participants are randomly divided into 2 groups. They will receive an 4 months lasting intervention in addition to the regular dance lessons. The time schedule of the intervention is identical for both groups. Participants from group A receive an active program aiming at improving their cardiovascular endurance, muscular strength and motor control. The level for cardiovascular training is based on the results of the maximal exercise test performed during baseline assessment. The level of training is determined at a level of 70% of the predicted maximal heart rate and was increased every 6 weeks with 5%, ending at 85%. Heart rate will be monitored during the training.

Participants from group B will receive an alternative program, in which all active parts are replaced by passive interventions. Several education sessions will be given regarding different topics, such as stress management, nutrition, injuries, etc. In addition, also practical sessions well be held to practice massage, passive stretching, taping. The intervention will be supervised by physical therapists and master students in Physiotherapy, experienced in dancing, motor control and/or physical conditioning, and an attendance list will register the presence of the participants.

The injuries of the dancers will be registered during the intervention and during a 6 months follow up period.

ELIGIBILITY:
Inclusion Criteria:

* students enrolled in the Bachelor of Dance at the Royal Conservatoire, Artesis Hogeschool in Lier, Belgium

Exclusion Criteria:

* No full time enrollment

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Changes in Physical condition | Post intervention (6 months after baseline evaluation)
  The physical condition is tested using an incremental exercise test on an electronically braked bicycle ergometer with a graded increase in workload. Fatigue during test performance is monitored every minute with a Borg scale from 6 (no fatigue) to 20 (complete exhaustion). There is continuous monitoring of electrocardiographic and ventilatory variables such as ventilation rate, respiration rate, VCO2 and VO2

SECONDARY OUTCOMES:
changes in musculoskeletal injury incidence during the intervention | during intervervention (6 months after baseline)
  A standardized questionnaire is used to collect demographic information at baseline, and an injury registration form is used to assess musculoskeletal symptoms and injuries (Cumps et al., 2007). Using this injury registration form, information is gathered about the occurrence of the symptoms and injuries, the time loss and the medical diagnosis. This injury registration form has already been used in prospective epidemiology research in sportsmen (Cumps et al., 2007) and in dancers (Roussel et al., 2009).
changes in motor control | post intervention (6 months after baseline)
  Lumbo-pelvic movement control is assessed by evaluating the subjects' ability to control movement of the lumbo-pelvic region while performing simple movements in the hips. Four commonly used clinical tests, i.e. the Active Straight Leg Raising, Bent Knee Fall Out, Knee Lift Abdominal Test and Standing Bow are used in the present study for the evaluation of lumbo-pelvic movement control. The reliability of these tests has been described elsewhere (Roussel et al. 2009a).
Changes in functional evaluation during the intervention | Post intervention (6 months after baseline)
  The SF-36 is a generic instrument in which health-related quality of life is measured. The dance functional outcome questionnaire consists of two parts: daily activities and dance-related functionality. For every question there are six possible responses, ranging from 'excellent functionality' to 'poor functionality'. The DFOS has very good test-retest reliability for healthy professional dancers and is very sensitive to functional changes in the dancers (Bronner et al., 2007).
Changes in Functional evaluation during follow up | Folow up (till 18 months after baseline evaluation)
  The same questionnaires will further be collected during the follow up period (12 and 18 months after baseline assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie A Roussel, PhD, Principal Investigator — Artesis University College; Wilfried De BAcker, PhD, MD, Study Director — Universiteit Antwerpen
Locations (1):
- Artesis University College, Antwerp, Belgium

REFERENCES:
- [Derived] Roussel NA, Vissers D, Kuppens K, Fransen E, Truijen S, Nijs J, De Backer W. Effect of a physical conditioning versus health promotion intervention in dancers: a randomized controlled trial. Man Ther. 2014 Dec;19(6):562-8. doi: 10.1016/j.math.2014.05.008. Epub 2014 Jun 3. PMID 24951437